CLINICAL TRIAL: NCT02322372
Title: Comparison of Conventional Dose Spinal Anesthesia With Low-dose Spinal Anesthesia and Femoral Blockade Combination in Outpatient Knee Arthroscopy
Brief Title: Femoral Blockade and Low-dose Spinal Anesthesia in Outpatient Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Sanem Cakar Turhan, Specialist, Ankara University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 30/06/2014
Record Dates: First submitted 2014-12-13; First posted 2014-12-23 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Meniscus Lesion
Keywords: femoral blockade; bupivacaine
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group F (Active Comparator): Ultrasound-guided femoral blockade with 15 mL of bupivacaine 0.5% diluted in 15 mL saline was performed in supine position. Then the patient was turned to lateral decubitus position with the operated extremity on dependant position and intrathecal injection of heavy bupivacaine 1 mL (5 mg) was administered from L3-L4 intervertebral space at a rate of 1 mL/20 second.
  .
  Interventions: Drug: Femoral blockade
- Group S (Active Comparator): The patient was turned to lateral decubitus position with the operated extremity on dependant position and intrathecal injection of heavy bupivacaine 2 mL (10 mg) was administered from L3-L4 intervertebral space at a rate of 1 mL/20 second.
  Interventions: Drug: Intrathecal anesthesia

INTERVENTIONS:
Drug: Femoral blockade — Spinal anesthesia with heavy bupivacaine combined with femoral blockade with bupivacaine
  Other Names: Marcaine
  Arms: Group F
Drug: Intrathecal anesthesia — Spinal anesthesia with heavy bupivacaine
  Other Names: Marcaine
  Arms: Group S

SUMMARY:
The investigators of the current study aimed to evaluate the effect of spinal anesthesia with low dose bupivacaine combined with femoral blockade on duration of anesthesia and time of first analgesic requirement during postoperative period

DETAILED DESCRIPTION:
Fifty patients undergoing arthroscopic meniscus repair were included to the current study.

The patients were allocated to two groups as the spinal anesthesia with conventional dose of heavy bupivacaine or spinal anesthesia with low dose heavy bupivacaine combined with femoral blockade.

Blood pressures and heart rates were recorded at the beginning, at the 0th minute following femoral block, at the 0th minute and in two-minute intervals following spinal anesthesia for 20 minutes and in five-minute intervals till the end of surgery.

The sensorial block and motor block in both extremities were recorded in two-minute intervals following spinal anesthesia and in five-minute intervals till the end of surgery The time of sensorial blockade to reach T12, maximum level of sensorial blockade level and the time to reach maximum level of sensorial blockade and the time for regression of sensorial blockade to L2, the time for regression of motor blockade were recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients aged between 25-65 undergoing arthroscopic meniscus repair

Exclusion Criteria:

* Contraindications to regional anesthesia (coagulopathy, severe aortic stenosis, sever mitral stenosis, increased intracranial pressure, severe hypovolemia, presence of infection on the site of injection)
* Presence of previous spinal surgery
* Presence of diabetes mellitus
* Presence of neurological disturbance
* Uncooperated patients, patients not accepting to participate the study
* Allergy to study drugs
* ASA II-IV patients, BMI >38, Height < 150 cm and >190 cm

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time of sensorial block to regress L2 | 24 hours

SECONDARY OUTCOMES:
Time of first analgesic requirement | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Akmese, Specialist, Principal Investigator — Ankara University Faculty of Medicine; Fatma Ozkan, Assistant, Principal Investigator — Ankara University Faculty of Medicine
Locations (1):
- Ankara University Medical School Anesthesiology and ICU Department, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Turhan KS, Akmese R, Ozkan F, Okten FF. Comparison of low-dose spinal anesthesia and single-shot femoral block combination with conventional dose spinal anesthesia in outpatient arthroscopic meniscus repair. Eur Rev Med Pharmacol Sci. 2015 Apr;19(8):1489-97. PMID 25967725